CLINICAL TRIAL: NCT03594708
Title: Impact of Immunonutrition Supplementation Combining Fermentable Fiber, Omega-3 Fatty Acids, Vitamin D, Vitamin E, and Zinc on Intestinal Inflammation, Gut Microbial Activity, and Severity of Symptoms in Ulcerative Colitis Patients
Brief Title: Immunonutrition in Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baptist Memorial Health Care Corporation (Other)
Responsible Party: Principal Investigator, Katherine Cook, Research Assistant, Baptist Memorial Health Care Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCS2018
Record Dates: First submitted 2018-01-19; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo consisting of rice starch, light olive oil, and vegetable oil
  Interventions: Dietary Supplement: Placebo supplement
- Supplement (Active Comparator): active supplement consisting of a fermentable fiber, omega-3 polyunsaturated fatty acid, vitamin D3, vitamin E, and zinc
  Interventions: Dietary Supplement: Nutrition supplement

INTERVENTIONS:
Dietary Supplement: Nutrition supplement — Fermentable fiber, omega-3 fatty acid, vitamin D3, vitamin E, zinc
  Arms: Supplement
Dietary Supplement: Placebo supplement — rice starch, light olive oil, vegetable oil
  Arms: Placebo

SUMMARY:
This study tests the hypothesis that a supplement that combines a functional fiber, long chain omega-3 polyunsaturated fatty acids (PUFAs), vitamin D3, vitamin E, and zinc will reduce clinical symptoms, decrease pro-inflammatory cytokines in the blood and ergo decrease inflammation, promote beneficial microbial activity in the colon, and help recovery of the intestinal mucosa of ulcerative colitis (UC) patients compared with a placebo.

DETAILED DESCRIPTION:
An anticipated 30 participants with newly diagnosed active ulcerative colitis will be recruited to participate in a randomized control trial, with 50% of the subjects distributed to the supplement (n=15) and the other 50% provided a placebo control (n=15). This is considered as a "proof of concept" study to determine if there is evidence that a multi-ingredient supplement (immunonutrition) will reduce UC disease severity.

ELIGIBILITY:
Inclusion Criteria:

* patients with active ulcerative colitis (proof of diagnosis from gastroenterologist), over 18 years old, has over 50% gut remaining, fully connected bowels (no colostomy), currently on 5-aminosalicylates (ASA) drugs, not pregnant or lactating

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduced inflammatory cytokines | 2 months
  cytokines will be isolated from blood analysis

SECONDARY OUTCOMES:
Improved microbiome/ increased Short-Chain Fatty acid (SCFA) counts | 2 months
  SCFA will be isolated from stool sample. SCFAs are anti-inflammatory components generated in the colon. The SCFAs looked at include acetate, lactate, propionate, butyrate, and isobutyrate.
Reduced bowel movements per day | 2 months
  Many with Ulcerative colitis can experience 10+ bowel movements per day. This intervention is aiming to reduce the total number of bowel movements per day
Decreased intestinal cramping/ pain | 2 months
  Many with ulcerative colitis experience constant intestinal cramping. This intervention is geared towards reducing pain and discomfort for the participants

CONTACTS AND LOCATIONS:
Overall Officials: Randal K Buddington, PhD, Principal Investigator — The University of Memphis
Locations (1):
- GI Specialists Foundation, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres MI, Rios A. Current view of the immunopathogenesis in inflammatory bowel disease and its implications for therapy. World J Gastroenterol. 2008 Apr 7;14(13):1972-80. doi: 10.3748/wjg.14.1972. PMID 18395894
- [Background] Lewis JD, Abreu MT. Diet as a Trigger or Therapy for Inflammatory Bowel Diseases. Gastroenterology. 2017 Feb;152(2):398-414.e6. doi: 10.1053/j.gastro.2016.10.019. Epub 2016 Oct 25. PMID 27793606
- [Background] Ruemmele FM. Role of Diet in Inflammatory Bowel Disease. Ann Nutr Metab. 2016;68 Suppl 1:33-41. doi: 10.1159/000445392. Epub 2016 Jun 30. PMID 27355913
- [Background] Rampertab S, Brown A. Inflammatory bowel disease. In: The Health Professional's Guide to Gastrointestinal Nutrition. Academy of Nutrition and Dietetics, 2015.
- [Background] Seidner DL, Lashner BA, Brzezinski A, Banks PL, Goldblum J, Fiocchi C, Katz J, Lichtenstein GR, Anton PA, Kam LY, Garleb KA, Demichele SJ. An oral supplement enriched with fish oil, soluble fiber, and antioxidants for corticosteroid sparing in ulcerative colitis: a randomized, controlled trial. Clin Gastroenterol Hepatol. 2005 Apr;3(4):358-69. doi: 10.1016/s1542-3565(04)00672-x. PMID 15822041